CLINICAL TRIAL: NCT04911075
Title: Depth of Necrosis in Normal Cervical Epithelium After 85% Trichloroacetic Acid (TCA) Application
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Dr Cipto Mangunkusumo General Hospital (Other)
Responsible Party: Principal Investigator, Prof. Dr. dr. Laila Nuranna, SpOG-K, Professor, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21020134
Record Dates: First submitted 2021-05-24; First posted 2021-06-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Cervix; Intraepithelial Neoplasia
Keywords: Trichloroacetic Acid (TCA); Depth of Necrosis; Cervix Intraepithelial Neoplasia
MeSH Terms: conditions — Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 85% TCA Group (Experimental): * Participants are subject who will undergo an elective total hysterectomy procedure for indications of gynecological organ abnormalities, whether benign, pre-cancerous, or malignant other than cervical pathology.
  * The 85 percent TCA solution will be applied to participants cervical tissue 24 hours before surgery.
  Interventions: Drug: 85% TCA Solution

INTERVENTIONS:
Drug: 85% TCA Solution — * TCA is an acetic acid analogue solution (CCl3COOH) which is formed from the reaction of acetic acid (CH3COOH) with chlorine (3Cl2).
  * High concentrations (85 percent) of this solution can penetrate deeply into the epidermis-dermis layer and cause cells necrosis.
  * This solution (1-2 milliliter) will be applied to participants cervical tissue (ectocervix and endocervix) using cotton swab for 1-3 minutes.
  Other Names: CCl₃COOH

SUMMARY:
Early detection and treatment of precancerous lesions are the pillars of cervical cancer prevention. Cervical Intraepithelial Neoplasia (CIN) is a precancerous lesion that histologically can be found in one of three stages of development; CIN-I (low grade), CIN-II, or CIN-III (collectively called high grade), depending on the proportion of the depth of the lesion to the thickness of the cervical epithelium. The higher the degree of CIN, the deeper the pre-cancerous lesions are found in the epithelial lining of the cervix. Therefore, from the point of view of precancerous lesions treatment, its effectiveness will be determined by the ability to eradicate all high-grade lesions. In other words, it has an effect that can reach depths beyond the depth of the high grade lesion.

According to a study in the US (1982), as many as 99.7% of CIN-III cases had a lesion depth of less than 4.8 millimeter. Furthermore, a Netherlands study (1990) stated that as many as 99.7% of CIN-III cases had a maximum lesion depth of 3.6 millimeters. While in subjects from developing countries, study from Peru (2018) showed that 93.5% of CIN-III cases have a lesion depth of less than 5 millimeters. Based on the results of these studies, a treatment for CIN can only be said to be effective if it can create a therapeutic effect which can reach depths of 4-5 millimeters in cervix epithelial.

Trichloroacetic acid (TCA) is an acetic acid analogue, which has long been known as a chemical peel and also frequently used to treat genital ward and precancerous skin lesions. The effect of TCA therapy is the destruction of the epithelium forming epithelial necrosis, followed by re-epithelialization of the supporting tissue and stimulation of collagen synthesis within approximately in 24 hours. There are no studies regarding the depth of cervical necrosis that can be achieved by application of this solution to the cervix epithelial.

DETAILED DESCRIPTION:
Primary Objectives:

The purpose of this study is to determine the depth of epithelial necrosis in cervical tissue specimen after 85 percent TCA application on clinically normal cervix.

Procedure:

Patients will receive a single administration of 1-2 milliliter of 85 percent TCA in 24 hours before elective total hysterectomy surgery on indication other than cervical pathology. The 85 percent TCA will be applied topically onto the ectocervix and the endocervix canal with a cotton swab for 1-2 minutes. After surgery, cervical specimen will be fixated in formalin and sent for histopathologic examination.

ELIGIBILITY:
Inclusion Criteria:

* Normal cervix without significant changes and must be tested negative for Visual Inspection Acetic-Acid (VIA) test (no acetowhite lesions are found)
* Participants are willing to participate voluntarily in this research by signing a consent form.

Exclusion Criteria:

* Patients who finally have undergone sub-total or supra-vaginal hysterectomy.
* Any abnormalities found in postoperative cervical histopathology results.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-04-15 (Actual); Primary Completion 2021-10-25 (Actual); Study Completion 2021-10-25 (Actual)

PRIMARY OUTCOMES:
Depth of Cervical Epithelial Ablation | 30 days
  Based on damage to the cervical epithelium, both squamous (ectocervix), transformation zone, and columnar (endocervix) epithelium. Destruction of base membrane and stromal tissue will also be evaluated. Microscopic evaluation using a micrometer on a 10 times magnification eyepiece. The deepest ablative destruction in epithelial, base membrane, and stromal tissue will be recorded and stated in millimetres.

SECONDARY OUTCOMES:
Pain Scores | 10 minutes
  Measured immediately after application of the 85 percent TCA solution with Visual Analogue Scale (VAS) score. Highest score means worse ouctcome. Minimum score is 0 (No Pain) and maximum score is 10 (worst pain).

CONTACTS AND LOCATIONS:
Overall Officials: Laila Nuranna, Professor, Principal Investigator — Indonesia University
Locations (1):
- dr. Cipto Mangunkusumo National Central General Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Yes
All Individual Patient Data (IPD) that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: IPD will become available 1 year after publication for duration of 1 year
Access Criteria: IPD will be shared with investigators from Indonesia and any additional supporting information will be shared, including with whom, for what types of analyses, and by what mechanism. Information about who will review requests and criteria for reviewing requests may also be provided.

REFERENCES:
- [Background] Boonstra H, Aalders JG, Koudstaal J, Oosterhuis JW, Janssens J. Minimum extension and appropriate topographic position of tissue destruction for treatment of cervical intraepithelial neoplasia. Obstet Gynecol. 1990 Feb;75(2):227-31. PMID 2300349
- [Background] Abdul-Karim FW, Fu YS, Reagan JW, Wentz WB. Morphometric study of intraepithelial neoplasia of the uterine cervix. Obstet Gynecol. 1982 Aug;60(2):210-4. PMID 7155483
- [Background] Taxa L, Jeronimo J, Alonzo TA, Gage J, Castle PE, Cremer ML, Felix JC. Depth of Cervical Intraepithelial Neoplasia Grade 3 in Peruvian Women: Implications for Therapeutic Depth of Necrosis. J Low Genit Tract Dis. 2018 Jan;22(1):27-30. doi: 10.1097/LGT.0000000000000355. PMID 29271853
- [Background] Brodland DG, Cullimore KC, Roenigk RK, Gibson LE. Depths of chemexfoliation induced by various concentrations and application techniques of trichloroacetic acid in a porcine model. J Dermatol Surg Oncol. 1989 Sep;15(9):967-71. doi: 10.1111/j.1524-4725.1989.tb03183.x. PMID 2778185
- [Background] Mariategui J, Santos C, Taxa L, Jeronimo J, Castle PE. Comparison of depth of necrosis achieved by CO2- and N2O-cryotherapy. Int J Gynaecol Obstet. 2008 Jan;100(1):24-6. doi: 10.1016/j.ijgo.2007.07.009. Epub 2007 Sep 25. PMID 17897647
- [Background] Adepiti AC, Ajenifuja OK, Fadahunsi OO, Osasan SA, Pelemo OE, Loto MO. Comparison of the depth of tissue necrosis between double-freeze and single-freeze nitrous oxide-based cryotherapy. Niger Med J. 2016 Jan-Feb;57(1):1-4. doi: 10.4103/0300-1652.180561. PMID 27185971
- [Background] Geisler S, Speiser S, Speiser L, Heinze G, Rosenthal A, Speiser P. Short-Term Efficacy of Trichloroacetic Acid in the Treatment of Cervical Intraepithelial Neoplasia. Obstet Gynecol. 2016 Feb;127(2):353-9. doi: 10.1097/AOG.0000000000001244. PMID 26942365
- [Background] Walker DC, Brown BH, Blackett AD, Tidy J, Smallwood RH. A study of the morphological parameters of cervical squamous epithelium. Physiol Meas. 2003 Feb;24(1):121-35. doi: 10.1088/0967-3334/24/1/309. PMID 12636191

DOCUMENTS (2):
  • Statistical Analysis Plan (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04911075/SAP_000.pdf
  • Informed Consent Form (2021-02-15): https://cdn.clinicaltrials.gov/large-docs/75/NCT04911075/ICF_001.pdf